CLINICAL TRIAL: NCT05683535
Title: Adverse Events Questionnaire for Low Dose Atropine Eye Drops
Brief Title: Adverse Events Related to Low Dose Atropine
Acronym: AELDA
Status: Completed | Type: Observational
Sponsor: Scripps Health (Other)
Responsible Party: Sponsor
Other Study IDs: AELDA
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Myopia, Progressive
Keywords: adverse events; nearsightedness; atropine
MeSH Terms: conditions — Myopia, Degenerative; Myopia | interventions — Atropine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Atropine Sulfate — 0.01%, 0.03%, or 0.05% atropine eye drops made from compounding pharmacies.

SUMMARY:
Progressive myopia can lead to severe vision loss and is associated with retinal detachment, glaucoma, and other comorbidities. Several studies have shown that off-label, low-dose atropine eye drops slow the progression of myopia. Many eye care providers are now prescribing off-label atropine eye drops for their myopic patients, with the prescribed concentrations varying amongst providers.

The purpose of this study is to determine if low-dose atropine eyedrops used daily, cause adverse effects to the eyes. Patients currently using 0.01%, 0.03%, or 0.05% atropine eye drops obtained from compounding pharmacies will be assessed for associated adverse effects.

DETAILED DESCRIPTION:
Eligibility: Myopic patients currently using 0.01%, 0.03%, or 0.05% atropine eye drops, prescribed by the investigator(s).

Patients that meet the eligibility criteria will be given the parental consent form and child assent form (if applicable) during their regularly scheduled office visit. After consent forms are signed and at each follow-up visit, the investigator or study coordinator will begin by querying for adverse events by asking each patient general, non-directed questions, such as "How have you been feeling since the last visit?" Directed questioning and examination will then be done as appropriate. All reported adverse events will be documented on the appropriate CRF. The patients will then continue with their regular eye exam.

Patients enrolled in the study will be assessed for adverse events at each regularly scheduled office visit for the duration of the study (up to 5 years), unless they choose to withdraw from the study.

The study will assess 148 patients using either 0.01%, 0.03%, or 0.05% atropine eye drops (prescribed by the investigator), over a five-year period.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with myopia
* patients must be currently using 0.01%, 0.03%, or 0.05% atropine eye drops daily
* low-dose atropine eye drops must be prescribed by the principal investigator and obtained from a compounding pharmacy

Exclusion Criteria:

* patients without myopia
* patients with myopia, but not using low-dose atropine eye drops

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric patients diagnosed with myopia and using either 0.01%, 0.03%, or 0.05% atropine eye drops daily, prescribed by the principal investigator.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Summary of adverse events by dose level at the time of the adverse event | up to 5 years
  Summary of total adverse events and severity of adverse events, by dose level at time of the adverse event

OTHER OUTCOMES:
Summary of Source of Atropine | up to 5 years
  Summary of name of compounding pharmacy, cost of eye drops, size of the bottle of eye drops, and if there was a delay in obtaining eye drops from the compounding pharmacy.
Summary of adverse events by starting dose | up to 5 years
  Summary of adverse events by dose of atropine prescribed at start of study
Summary of demographics and medical history by atropine starting dose | up to 5 years
  Summary of demographics and medical history by atropine starting dose

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Ostrow, MD, Principal Investigator — Scripps Health
Locations (1):
- Laura Kirkeby, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leo SW; Scientific Bureau of World Society of Paediatric Ophthalmology and Strabismus (WSPOS). Current approaches to myopia control. Curr Opin Ophthalmol. 2017 May;28(3):267-275. doi: 10.1097/ICU.0000000000000367. PMID 28212157
- [Background] Gong Q, Janowski M, Luo M, Wei H, Chen B, Yang G, Liu L. Efficacy and Adverse Effects of Atropine in Childhood Myopia: A Meta-analysis. JAMA Ophthalmol. 2017 Jun 1;135(6):624-630. doi: 10.1001/jamaophthalmol.2017.1091. PMID 28494063
- [Background] Pineles SL, Kraker RT, VanderVeen DK, Hutchinson AK, Galvin JA, Wilson LB, Lambert SR. Atropine for the Prevention of Myopia Progression in Children: A Report by the American Academy of Ophthalmology. Ophthalmology. 2017 Dec;124(12):1857-1866. doi: 10.1016/j.ophtha.2017.05.032. Epub 2017 Jun 29. PMID 28669492
- [Background] Chia A, Chua WH, Cheung YB, Wong WL, Lingham A, Fong A, Tan D. Atropine for the treatment of childhood myopia: safety and efficacy of 0.5%, 0.1%, and 0.01% doses (Atropine for the Treatment of Myopia 2). Ophthalmology. 2012 Feb;119(2):347-54. doi: 10.1016/j.ophtha.2011.07.031. Epub 2011 Oct 2. PMID 21963266
- [Background] Yam JC, Jiang Y, Tang SM, Law AKP, Chan JJ, Wong E, Ko ST, Young AL, Tham CC, Chen LJ, Pang CP. Low-Concentration Atropine for Myopia Progression (LAMP) Study: A Randomized, Double-Blinded, Placebo-Controlled Trial of 0.05%, 0.025%, and 0.01% Atropine Eye Drops in Myopia Control. Ophthalmology. 2019 Jan;126(1):113-124. doi: 10.1016/j.ophtha.2018.05.029. Epub 2018 Jul 6. PMID 30514630
- [Background] Fu A, Stapleton F, Wei L, Wang W, Zhao B, Watt K, Ji N, Lyu Y. Effect of low-dose atropine on myopia progression, pupil diameter and accommodative amplitude: low-dose atropine and myopia progression. Br J Ophthalmol. 2020 Nov;104(11):1535-1541. doi: 10.1136/bjophthalmol-2019-315440. Epub 2020 Feb 21. PMID 32086237
- [Background] Chia A, Lu QS, Tan D. Five-Year Clinical Trial on Atropine for the Treatment of Myopia 2: Myopia Control with Atropine 0.01% Eyedrops. Ophthalmology. 2016 Feb;123(2):391-399. doi: 10.1016/j.ophtha.2015.07.004. Epub 2015 Aug 11. PMID 26271839
- [Background] Chia A, Chua WH, Wen L, Fong A, Goon YY, Tan D. Atropine for the treatment of childhood myopia: changes after stopping atropine 0.01%, 0.1% and 0.5%. Am J Ophthalmol. 2014 Feb;157(2):451-457.e1. doi: 10.1016/j.ajo.2013.09.020. Epub 2013 Dec 4. PMID 24315293
- [Background] Yam JC, Li FF, Zhang X, Tang SM, Yip BHK, Kam KW, Ko ST, Young AL, Tham CC, Chen LJ, Pang CP. Two-Year Clinical Trial of the Low-Concentration Atropine for Myopia Progression (LAMP) Study: Phase 2 Report. Ophthalmology. 2020 Jul;127(7):910-919. doi: 10.1016/j.ophtha.2019.12.011. Epub 2019 Dec 21. PMID 32019700
- [Background] Chua WH, Balakrishnan V, Chan YH, Tong L, Ling Y, Quah BL, Tan D. Atropine for the treatment of childhood myopia. Ophthalmology. 2006 Dec;113(12):2285-91. doi: 10.1016/j.ophtha.2006.05.062. Epub 2006 Sep 25. PMID 16996612